CLINICAL TRIAL: NCT05978115
Title: Clinical and Radiographic Evaluation of Three Different Modalities for Management of Distal Extension Atrophied Mandibular Ridge: A One Year Prospective Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Mohamed shady, Assistant Professor, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: A01020822
Record Dates: First submitted 2023-07-28; First posted 2023-08-07 (Actual); Last update posted 2023-08-07 (Actual); Status verified 2023-07

CONDITIONS: Different Treatment Outcomes of Atrophied Distal Extension Cases
MeSH Terms: interventions — Dental Prosthesis, Implant-Supported

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- short implant supported removable partial overdenture (Experimental)
  Interventions: Procedure: implant supported prosthesis
- short Implant supported fixed partial denture (Experimental)
  Interventions: Procedure: implant supported prosthesis
- Ridge Augmentation and implant supported fixed partial denture (Experimental)
  Interventions: Procedure: implant supported prosthesis

INTERVENTIONS:
Procedure: implant supported prosthesis — Group A: short dental implant placement + Removable partial denture Group B: Short implant placement + Fixed partial denture Group c: Bone Augmentation + Implant placement + Fixed Partial denture
  Other Names: Bone augmentation for atrophied ridge

SUMMARY:
Nine patients selected for this study with mandibular free end saddle and atrophied posterior ridge according to treatment options all patients will be divided randomly into 3 groups:

* Group A: included three participants who will receive implant retained partial overdentures
* Group B: included three participants who will receive short implants supported fixed prosthesis
* Group C: included three participants who will receive long implant supported fixed prosthesis after ridge augmentation.
* For Group A: Implant retained partial overdenture The implants will be inserted in first premolar areas and partial overdenture will be connected with implant by locator attachment.
* For Group B: Short implant supported fixed prosthesis The implants will be inserted in first premolar, second premolar, and first molar areas without any ridge augmentation and the implant will be connected by fixed prosthesis
* For group C: Long implant supported fixed prosthesis after ridge augmentation The implants will be inserted in first premolar, second premolar, and first molar areas with ridge augmentation by using Khoury technique17 and the implants will be connected by fixed prosthesis
* Clinical evaluation will be made in terms of:

  * Gingival Index (GI)
  * Plaque Index (PI)
  * Pocket Depth (PD)
  * Width of Keratinized Mucosa (KM)
  * Implant Stability (ISQ).
* Radiographic evaluation will include mandibular residual ridge resorption using the proportional area measurements.

evaluation periods will be performed at time of insertion T(0), 6 months after insertion T(6), 12 months after insertion T(6)

DETAILED DESCRIPTION:
Introduction Long span distal-extension removable partial dentures (RPDs) are associated with several problems related to their stability, retention, esthetics, and masticatory efficiency.1,2 The lack of distal dental support in mandibular Kennedy class I distal extension-RPDs results in transmission of vertical, horizontal, and torsional forces to supporting tissues during mastication with subsequent adverse changes in both abutment teeth and edentulous areas. In addition, constant pressure from the denture base gradually causes ridge resorption under the denture base.3-5 Prosthodontic management of long span distal extension partially edentulous patients has expanded with the introduction of Osseo integrated implants.6 The use of implants to support and retain distal extension partial overdentures has been reported to minimize RPD dislodgement, provide additional retention and stability, prevent the development of combination syndrome and improve patient satisfaction in a cost-effective manner.7,8 Moreover, placing bilateral dental implants distal to canine area of the residual alveolar ridges is becoming a popular treatment choice in case of limited height of posterior mandibular ridge7,9,10 Such prostheses can be retained to the implants with different unsplinted anchors such as ball, Locator, and magnetic attachments.1 Although Implant-supported distal extension prosthesis could be an ideal treatment option, alveolar resorption, lack of sufficient bone volume and proximity to the inferior alveolar nerve, presenting a difficult clinical situation for positioning endosseous implants. A bone height of 10-12mm is generally considered to be the minimal amount of bone required to place implants of ''sufficient'' length, 9-11mm long, which are most likely to generate good long-term results and to minimize the risk of permanent damage to the alveolar inferior nerve.11 Often times, however, the amount of residual bone above the mandibular canal is <10mm, and implant placement is considered at a higher risk of failure.11To address a case of reduced bone height in the posterior mandible, either ridge augmentation or placement of short implant could be the proposed approaches.

The development of bone augmentation procedures has allowed placement of dental implants into jawbone areas lacking an amount of bone sufficient for standard implant placement.11 While augmentation procedures can yield favorable outcomes, they can be associated with significant postoperative morbidity and complications.12 On the other hand, short implants could be a simpler, cheaper, and faster alternative to augmentation procedures, even if in some "critical cases" the residual bone crest above the inferior alveolar nerve is only 5-7 mm in height, and therefore the surgical augmentation treatment is mandatory.11,12 However, it is commonly perceived that short implants do not have a good long-term prognosis when compared with longer implants. Although preliminary findings suggest that short implants may be a better alternative to various bone augmentation procedures, long-term follow-up evaluations are indicated to draw definitive conclusion.13-15 Implant-supported removable prostheses improve patients' satisfaction with treatment and quality of life. When canines are the only present abutments, insertion of the implants distal the canine areas can provide support and retention, eliminate the use of unesthetic retentive clasps, and prevent unfavorable horizontal forces that may damage the abutment periodontium. However, some biological and mechanical complications remain. Mechanical complications associated with implant-supported overdentures are loss of retention of attachment systems, the need to replace retention elements and to reline or repair the resin portion of the denture, and implant fracture. Despite their success, implant-supported removable prostheses require periodic maintenance.

Based on the proceeding, three treatment modalities could be the solution for long span distal-extension removable partial dentures (RPDs); implant retained partial overdenture, short implant supported fixed prosthesis, and long implant supported fixed prosthesis after ridge augmentation. Comparing the clinical and radiographic outcomes of the three different treatment modalities are relatively scarce in literature to explore which treatment is more appropriate regarding periodontal tissue health and patient satisfaction.

Aim of the work This study will aim to assess the clinical and radiographic outcomes of three different treatments modalities for management of distal extension atrophied mandibular ridge; A; implant retained partial overdenture, B; short implant supported fixed prosthesis, C; long implant supported prosthesis after ridge augmentation

* Clinical evaluation will be made in terms of:

  • Gingival Index (GI)

  • Plaque Index (PI)
  * Pocket Depth (PD)
  * Width of Keratinized Mucosa (KM)
  * Implant Stability (ISQ).
* Radiographic evaluation will include mandibular residual ridge resorption using the proportional area measurements.

Materials and Methods

1. Patient selection and grouping:

Nine patients aged between (45 to 70 years) will be selected from outpatient clinic of the Removable Prosthodontic Department, Faculty of Dentistry, Mansoura University, Egypt.

* All selected participants will be required to have the following inclusion criteria:

  1. Atrophied partially edentulism in the posterior mandible having a residual bone height of 6-8mm bone between inferior alveolar nerve and crest of the ridge to receive implants 2. Residual alveolar ridges covered with healthy mucosa without any signs of inflammation or remaining roots.

  3. Normal maxilla-mandibular relationship with sufficient available restorative space.16
* Patients with the following conditions will be excluded:

  1. Diseases that affect bone metabolism, eg: uncontrolled diabetes, hyperparathyroidism, and osteoporosis.
  2. Systemic diseases that may affect osteointegration or complicate surgical procedures, eg: liver diseases, heart diseases and radiotherapy in head and neck region.
  3. Abnormal or harmful habits eg: smoking, bruxism, and clenching.
  4. Uncooperative patients and patients with poor oral hygiene.
* The study protocol will be reviewed and approved by ethical committee of the Faculty of Dentistry, Mansoura University
* Detailed written information about treatment strategy will be provided to all participants who meet the criteria, and then they will sign an informed consent. After consent will be given, eligible participants will be randomly divided into three groups:

  1. Group A: included three participants who will receive implant retained partial overdentures 2. Group B: included three participants who will receive short implants supported fixed prosthesis 3. Group C: included three participants who will receive long implant supported fixed prosthesis after ridge augmentation.

  2. Surgical and prosthetic procedures:
* Cone Beam Computed Tomography (CBCT) will be performed for each patient to mark implant placement sites, detect magnification errors, and select proper implant lengths. The implants will be inserted using non-submerged flapless surgical approach with the same operator in all groups.
* For Group A: Implant retained partial overdenture The implants will be inserted in first premolar areas and partial overdenture will be connected with implant by locator attachment.
* For Group B: Short implant supported fixed prosthesis The implants will be inserted in first premolar, second premolar, and first molar areas without any ridge augmentation and the implant will be connected by fixed prosthesis
* For group C: Long implant supported fixed prosthesis after ridge augmentation The implants will be inserted in first premolar, second premolar, and first molar areas with ridge augmentation by using Khoury technique17 and the implants will be connected by fixed prosthesis

  3. Evaluation of peri-implant tissues Clinical and radiographic evaluations of peri-implant tissues will be performed after definite prosthesis insertion (T0), six (T6) and twelve (T12) months after insertion.

A. Clinical evaluation

* The parameters for clinical evaluation of peri-implant tissue included: plaque index, gingival index, pocket depth, thickness of keratinized mucosa, and implant stability.

  1. Gingival index (GI):

     Modified gingival index will be recorded according to Mombelli et al.18, as follows: score 0; normal gingival, score 1; mild inflammation (slight change in color & slight edema), but no bleeding on probing, score 2; moderate inflammation (redness & edema), and bleeding on probing, and score 3; sever inflammation (marked redness, edema & ulceration) with tendency to spontaneous bleeding.
  2. Plaque index (PI):

     Plaque will be assessed according to modified plaque index describe by Mombelli et al.18 as follows: score 0; no plaque detected, score 1; plaque recognized only by running a probe across a smooth marginal surface of the implant, score 2; plaque can be seen by naked eye, and score 3; abundance of soft mater.
  3. Pocket depth (PD):

     Using a calibrated plastic periodontal probe, the distance between marginal border of the gingiva and the tip of the probe will be measured in mm and considered as pocket depth (PD).19
  4. The width of keratinized mucosa (KM):

     The width of peri-implant keratinized mucosa will be measured in mm using a calibrated plastic periodontal probe. Differences in color, texture and mobility between the keratinized mucosa and the lining mucosa served as markers for the detection of the muco-gingival junction.20 KM was then measured as the distance between the gingival margin and the muco-gingival junction.
  5. Implant stability (ISQ):
* Implant stability will be assessed using resonance frequency analysis (RFA). The resonance frequencies will be measured with the osstell® device (implant stability meter) and expressed with ISQ measurement scale (implant stability quotient). 21,22

B. Radiographic evaluation:

* Radiographic evaluation will be assessed using Cone Beam Computed Tomography (CBCT) and periapical radiographic X ray.
* Implant dimensions in the radiographs will be compared with actual implant dimensions to detect magnification errors. The ratio between implant dimensions in the radiographs and actual implant dimensions will be used to modify the apparent measurement of peri-implant bone levels in the radiographs to obtain their actual values.
* Crestal alveolar bone changes will be determined along vertical and horizontal planes as recommended by Elsyad et al. 19,23
* For vertical alveolar bone changes: the distance between implant shoulder (A point) and first bone to implant contact (B point) called DIB, indicates vertical bone level in mm (AB line)
* For horizontal alveolar bone changes: the distance between the marginal bone level (C point) [ which represents the intersection point of a tangent to the horizontal bone crest (CD line) and another tangent to the crater-shaped defect (CB line)] and the implant perpendicularly: indicates horizontal bone level(mm).
* Vertical bone loss (VBL) will be calculated by subtracting DIB at T6 and T12 from DIB at T0. Horizontal bone loss (HBLO) will be calculated by subtracting HBL at T6 and T12 from HBL at T0.
* Crestal alveolar bone changes (vertical and horizontal bone loss) will be measured at mesial and distal surface of each implant.

C. Implant survival To estimate the cumulative survival rate, a Kaplan-Meier analysis will be used, involving the following clinical parameters for success suggested by Albrektsson and Isidor 24; no clinical problems (pus, suppuration, implant mobility and pain) and limited change in peri-implant crestal bone level, as assessed by radiographic follow-up: during the first year of loading ≤ 1.5 mm and annual additional bone loss thereafter ≤ 0.2 mm/year. An implant was classified as a 'survived implant' when it was still functioning, irrespective of its conditions and do not need immediate removal, but did not fulfill the success criteria.

ELIGIBILITY:
Inclusion Criteria:

* All selected participants will be required to have the following inclusion criteria:

  1. Atrophied partially edentulism in the posterior mandible having a residual bone height of 6-8mm bone between inferior alveolar nerve and crest of the ridge to receive implants
  2. Residual alveolar ridges covered with healthy mucosa without any signs of inflammation or remaining roots.
  3. Normal maxilla-mandibular relationship with sufficient available restorative space.

Exclusion Criteria:

* -Patients with the following conditions will be excluded:

  1. Diseases that affect bone metabolism, eg: uncontrolled diabetes, hyperparathyroidism, and osteoporosis.
  2. Systemic diseases that may affect osteointegration or complicate surgical procedures, eg: liver diseases, heart diseases and radiotherapy in head and neck region.
  3. Abnormal or harmful habits eg: smoking, bruxism, and clenching.
  4. Uncooperative patients and patients with poor oral hygiene.

Ages: 50 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2021-08-20 (Actual); Primary Completion 2022-11-20 (Actual); Study Completion 2024-02-01 (Estimated)

PRIMARY OUTCOMES:
Gingival Index (GI) | at time of insertion of prosthesis T(0), 6 months after insertion T(6), 12 months after insertion T(12)
  Modified gingival index will be recorded according to Mombelli et al, as follows: score 0; normal gingival, score 1; mild inflammation (slight change in color & slight edema), but no bleeding on probing, score 2; moderate inflammation (redness & edema), and bleeding on probing, and score 3; sever inflammation (marked redness, edema & ulceration) with tendency to spontaneous bleeding.
Plaque Index (PI) | at time of insertion of prosthesis T(0), 6 months after insertion T(6), 12 months after insertion T(12)
  Plaque will be assessed according to modified plaque index describe by Mombelli et al. as follows: score 0; no plaque detected, score 1; plaque recognized only by running a probe across a smooth marginal surface of the implant, score 2; plaque can be seen by naked eye, and score 3; abundance of soft mater.
Pocket Depth (PD) | at time of insertion of prosthesis T(0), 6 months after insertion T(6), 12 months after insertion T(12)
  Using a calibrated plastic periodontal probe, the distance between marginal border of the gingiva and the tip of the probe will be measured in mm and considered as pocket depth (PD).
Width of Keratinized Mucosa (KM) | at time of insertion of prosthesis T(0), 6 months after insertion T(6), 12 months after insertion T(12)
  The width of peri-implant keratinized mucosa will be measured in mm using a calibrated plastic periodontal probe. Differences in color, texture and mobility between the keratinized mucosa and the lining mucosa served as markers for the detection of the muco-gingival junction. KM was then measured as the distance between the gingival margin and the muco-gingival junction.
Implant Stability (ISQ) | at time of insertion of prosthesis T(0), 6 months after insertion T(6), 12 months after insertion T(12)
  Implant stability will be assessed using resonance frequency analysis (RFA). The resonance frequencies will be measured with the osstell® device (implant stability meter) and expressed with ISQ measurement scale (implant stability quotient).

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Shady, MD, Principal Investigator — Mansoura University Faculty of Dentistry, Prosthodontics department
Locations (1):
- Mansoura University, Faculty of dentistry, Al Mansurah, Egypt

REFERENCES:
- [Derived] Raffat EM, Shady M, Elkashty AAR, Syad ME. Comparative analysis of implant survival, peri-implant health, and patient satisfaction among three treatment modalities in atrophic posterior mandibles: a randomized clinical study. BMC Oral Health. 2025 Jun 7;25(1):939. doi: 10.1186/s12903-025-06286-7. PMID 40483406